CLINICAL TRIAL: NCT05478902
Title: Effectiveness of Non-surgical Management in Rotator Cuff Calcific Tendinopathy: a Randomised Clinical Trial (THE EFFECT TRIAL)
Brief Title: Effectiveness of Non-surgical Management in Rotator Cuff Calcific Tendinopathy (THE EFFECT TRIAL)
Acronym: EFFECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Lirios Dueñas, PhD Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1718862
Record Dates: First submitted 2022-07-21; First posted 2022-07-28 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Rotator Cuff Tendinosis; Rotator Cuff Injuries; Shoulder Tendinitis; Calcific Shoulder Tendinitis; Calcification Tendon; Calcific Tendinitis; Shoulder Pain
Keywords: exercise therapy; lavage; rotator cuff calcific tendinopathy; shoulder calcification; extracorporeal shockwave therapy; ultrasound-guided percutaneous irrigation; shoulder pain; shape up my shoulders; sums
MeSH Terms: conditions — Rotator Cuff Injuries; Rotator Cuff Tear Arthropathy; Shoulder Pain | interventions — Exercise Therapy; Extracorporeal Shockwave Therapy; Therapeutic Irrigation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Exercise Therapy (Experimental): This group will receive the Shape Up My Shoulders (SUMS) protocol and it will be led by a physiotherapist trained in therapeutic exercise. It will last 12 weeks and it will be divided in 3 stages.
  Stage I- Early-stage rehabilitation exercises (i.e., breathing and relaxation exercises, ball rolling exercises, hand gripping exercises, mental imagery and contralateral side exercises) and Shoulder Symptom Modification Procedure (SSMP). This stage typically lasts 1 to 2 weeks.
  Stage II - Isometric, eccentric and heavy slow resistance exercises. The final part of Stage II is a progression from eccentric only to eccentric and concentric contractions.
  Stage III - Functional program. This stage starts in week 5 or 6 and progressed to week 12. Involves pushing, pulling, throwing, lifting, carrying, and precision (sensory-motor control) exercises.
  Interventions: Procedure: Exercise Therapy
- Extracorporeal Shockwave Therapy (Active Comparator): This group will receive high energy Extracorporeal Shockwave Therapy (ESWT) applied by an experienced physiotherapist. ESWT will be applied on the most tender point of the shoulder, located by palpation. The dose will be 1500 impulses per session without anaesthesia and an intensity between 0.15 and 0.30 mJ/mm2 depending on patient tolerance. A total of 4 treatment sessions (1 session per week) with 1 week of rest between sessions will be implemented. Patient's position during the treatment will be seated in supine position with shoulder hyperextension and internal rotation with the hand placed below the contralateral glute with the palm touching the table.
  Interventions: Procedure: Extracorporeal Shockwave Therapy
- Ultrasound-Guided Percutaneous Irrigation (Active Comparator): This intervention will be performed by an experienced interventionist radiologist in two sessions. The shoulder position will be with hyperextension and internal rotation with the hand behind the back. One 20 mL syringe with saline solution, one with an anaesthetic with 20 mg/mL of mepivacaine 2% and another syringe with a corticoid injection with 40 mg/mL of triamcinolone acetonide will be prepared before the intervention. Firstly, the anaesthetic will be injected directed to the calcification. Then, the procedure will consist of injecting saline solution and aspiring the calcific deposits until it is neither possible to aspire more inside the syringe nor to detect any calcifications with ultrasound imaging. After that, a corticoid will be injected to the bursa to prevent the appearance of subacromial bursitis. Finally, an anaesthetic will be injected during the extraction of the needle.
  Interventions: Procedure: Ultrasound-Guided Percutaneous Irrigation
- Wait and Watch group (No Intervention): The wait and see group will not receive any intervention and will serve as a control group to determine the natural history of RCCT. If one treatment proves to be more effective then participants in the other groups will be offered that treatment after 12 months, or before, if the investigation finishes early due to an obvious group difference and a need to break randomisation codes.

INTERVENTIONS:
Procedure: Exercise Therapy — Exercise protocol for rotator cuff related shoulder pain
  Other Names: Shape Up My Shoulders Protocol
  Arms: Exercise Therapy
Procedure: Extracorporeal Shockwave Therapy — High Energy Extracorporeal Shockwave Therapy
  Arms: Extracorporeal Shockwave Therapy
Procedure: Ultrasound-Guided Percutaneous Irrigation — Two sessions of Ultrasound-Guided Percutaneous Irrigation
  Other Names: Lavage
  Arms: Ultrasound-Guided Percutaneous Irrigation

SUMMARY:
The aim of this study will be to compare the effectiveness of an exercise therapy program with extracorporeal shockwave therapy, ultrasound-guided percutaneous irrigation and a wait and see approach in people with rotator cuff calcific tendinopathy.

DETAILED DESCRIPTION:
Rotator cuff calcific tendinopathy (RCCT) is a common musculoskeletal disorder caused by the presence of calcific deposits in the rotator cuff with an important impact in the quality of life of those who are suffering it. Conservative interventions such as extracorporeal shockwave therapy (ESWT) or ultrasound-guided percutaneous irrigation of calcific tendinopathy (US-PICT) have been commonly recommended as part of the early management for this clinical condition. Exercise therapy (ET) has shown to be an effective intervention for people with rotator cuff tendinopathy, but it has not been tested in people with RCCT yet. A randomised, single-blinded four parallel group clinical trial will be conducted. Participants (n=116) will be randomised in four groups: (1) ET; (2) ESWT; (3) US-PICT or (4) control.

ELIGIBILITY:
Inclusion Criteria:

* calcification deposit in the rotator cuff confirmed by diagnostic imaging (ultrasound, MRI or X-ray);
* pain and loss of function in the shoulder;
* not currently receiving physiotherapy or ESWT.

Exclusion Criteria:

* previous treatments on last year (e.g., injections, ESWT, US-PICT, surgery, etc.);
* other shoulder disorders or trauma (e.g., fractures, dislocations, rotator cuff tears, frozen shoulder or shoulder instability);
* known allergy to any of the pharmacological products used in the study;
* taking oral anticoagulants
* taking oral steroid within the six months prior to participation in the study;
* cancer, systemic disease, pregnancy or infection;
* neck pain.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Shoulder Pain And Disability Index (SPADI) | Baseline
  Pain and function shoulder scale. Patients are told to circle the number that best describes their pain where: 0 = no pain and 10 = the worst pain imaginable. The means of the two subscales are averaged to produce a total score ranging from 0 (best) to 100 (worst).
Shoulder Pain And Disability Index (SPADI) | 2 weeks
  Pain and function shoulder scale. Patients are told to circle the number that best describes their pain where: 0 = no pain and 10 = the worst pain imaginable. The means of the two subscales are averaged to produce a total score ranging from 0 (best) to 100 (worst).
Shoulder Pain And Disability Index (SPADI) | 4 months
  Pain and function shoulder scale. Patients are told to circle the number that best describes their pain where: 0 = no pain and 10 = the worst pain imaginable. The means of the two subscales are averaged to produce a total score ranging from 0 (best) to 100 (worst).
Shoulder Pain And Disability Index (SPADI) | 6 months
  Pain and function shoulder scale. Patients are told to circle the number that best describes their pain where: 0 = no pain and 10 = the worst pain imaginable. The means of the two subscales are averaged to produce a total score ranging from 0 (best) to 100 (worst).
Shoulder Pain And Disability Index (SPADI) | 12 months
  Pain and function shoulder scale. Patients are told to circle the number that best describes their pain where: 0 = no pain and 10 = the worst pain imaginable. The means of the two subscales are averaged to produce a total score ranging from 0 (best) to 100 (worst).

SECONDARY OUTCOMES:
Pain Intensity | Baseline
  Shoulder pain intensity reported by the patient will be assessed using a 100-mm visual analogue scale (VAS, 0-100, 0=minimum score, 100=maximum score). Higher values represent a better outcome (less pain). Flexion, abduction, external rotation and hand behind the back
Pain Intensity | 2 weeks
  Shoulder pain intensity reported by the patient will be assessed using a 100-mm visual analogue scale (VAS, 0-100, 0=minimum score, 100=maximum score). Higher values represent a better outcome (less pain). Flexion, abduction, external rotation and hand behind the back
Pain Intensity | 4 months
  Shoulder pain intensity reported by the patient will be assessed using a 100-mm visual analogue scale (VAS, 0-100, 0=minimum score, 100=maximum score). Higher values represent a better outcome (less pain). Flexion, abduction, external rotation and hand behind the back
Pain Intensity | 6 months
  Shoulder pain intensity reported by the patient will be assessed using a 100-mm visual analogue scale (VAS, 0-100, 0=minimum score, 100=maximum score). Higher values represent a better outcome (less pain). Flexion, abduction, external rotation and hand behind the back
Pain Intensity | 12 months
  Shoulder pain intensity reported by the patient will be assessed using a 100-mm visual analogue scale (VAS, 0-100, 0=minimum score, 100=maximum score). Higher values represent a better outcome (less pain). Flexion, abduction, external rotation and hand behind the back
Range of motion | Baseline
  Flexion, abduction and hand behind the back measured with a questionnaire with different stages. Degrees measured in different stages ranged from 0-30º, 30-60º, 60-90º, 90-120º, 120-150º and above 150º for flexion and abduction. For hand behind the back: hand to the hip, to the buttock, low back, mid back or between scapulas.
Range of motion | 4 months
  Flexion, abduction and hand behind the back measured with a questionnaire with different stages. Degrees measured in different stages ranged from 0-30º, 30-60º, 60-90º, 90-120º, 120-150º and above 150º for flexion and abduction. For hand behind the back: hand to the hip, to the buttock, low back, mid back or between scapulas.
Range of motion | 12 months
  Flexion, abduction and hand behind the back measured with a questionnaire with different stages. Degrees measured in different stages ranged from 0-30º, 30-60º, 60-90º, 90-120º, 120-150º and above 150º for flexion and abduction. For hand behind the back: hand to the hip, to the buttock, low back, mid back or between scapulas.
Type of calcification | Baseline
  according to the Gartner classification assessed with x-ray by an experienced radiologist
Type of calcification | 4 months
  according to the Gartner classification assessed with x-ray by an experienced radiologist
Type of calcification | 12 months
  according to the Gartner classification assessed with x-ray by an experienced radiologist
Size of the calcification | Baseline
  Measured in millimeters. Assessed with X-ray by an experienced radiologist
Size of the calcification | 4 months
  Measured in millimeters. Assessed with X-ray by an experienced radiologist
Size of the calcification | 12 months
  Measured in millimeters. Assessed with X-ray by an experienced radiologist
Location of the calcification | Baseline
  Which tendon is affected. Assessed with X-ray by an experienced radiologist
Location of the calcification | 4 months
  Which tendon is affected. Assessed with X-ray by an experienced radiologist
Location of the calcification | 12 months
  Which tendon is affected. Assessed with X-ray by an experienced radiologist
Morphology of the calcification | Baseline
  Isolated- fragmented - multiple. Assessed with X-ray by an experienced radiologist
Morphology of the calcification | 4 months
  Isolated-fragmented- multiple. Assessed with X-ray by an experienced radiologist
Morphology of the calcification | 12 months
  Isolated-fragmented- multiple. Assessed with X-ray by an experienced radiologist
Central Sensitization Inventory (CSI) | Baseline
  Patient-reported instrument to identify when patient's symptoms may be related to central sensitization
Pittsburgh Sleep Quality Index (PSQI) | Baseline
  Self-reported questionnaire for measuring the subjective perception of sleep quality
Fear Avoidance Beliefs Questionnaire (FABQ) | Baseline
  Patient-reported instrument for measuring fear avoidance and beliefs. The score range is 0 to 96, with a higher value reflecting a higher degree of fear avoidance beliefs.
Tampa Scale for Kinesiophobia (TSK) | Baseline
  Self-reported questionnaire for measuring fear of movement or fear of (re)injury
painDETECT Scale | Baseline
  Self-administered questionnaire, developed to quickly detect neuropathic pain, asking the patient about the pain experienced at the moment and with- in the last 4 weeks
Pain Catastrophizing Scale | Baseline
  Patient-reported outcome to measure catastrophization
EuroQoL-5D | Baseline
  Patient-reported outcome to measure quality of life
Hospital Anxiety and Depression Scale | Baseline
  Patient-reported outcome to measure psychological factors
Patient Satisfaction | 2 weeks
  Global impression of change
Patient Satisfaction | 4 months
  Global impression of change
Patient Satisfaction | 6 months
  Global impression of change
Patient Satisfaction | 12 months
  Global impression of change
Night Pain | Baseline
  How much has the pain affected the patient at night in the last 4 weeks. From 1 to 5. 5 means worst. 1: No pain. 2: Pain 1 or 2 nights in the last 4 weeks. 3: 1 or 2 nights a week. 4: Pain almost every night. 5: Pain every night.
Night Pain | 2 weeks
  How much has the pain affected the patient at night in the last 4 weeks. From 1 to 5. 5 means worst. 1: No pain. 2: Pain 1 or 2 nights in the last 4 weeks. 3: 1 or 2 nights a week. 4: Pain almost every night. 5: Pain every night.
Night Pain | 4 months
  How much has the pain affected the patient at night in the last 4 weeks. From 1 to 5. 5 means worst. 1: No pain. 2: Pain 1 or 2 nights in the last 4 weeks. 3: 1 or 2 nights a week. 4: Pain almost every night. 5: Pain every night.
Night Pain | 6 months
  How much has the pain affected the patient at night in the last 4 weeks. From 1 to 5. 5 means worst. 1: No pain. 2: Pain 1 or 2 nights in the last 4 weeks. 3: 1 or 2 nights a week. 4: Pain almost every night. 5: Pain every night.
Night Pain | 12 months
  How much has the pain affected the patient at night in the last 4 weeks. From 1 to 5. 5 means worst. 1: No pain. 2: Pain 1 or 2 nights in the last 4 weeks. 3: 1 or 2 nights a week. 4: Pain almost every night. 5: Pain every night.

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Lluch, PT, PhD, Study Director — University of Valencia
Locations (2):
- Spain (2):
  - Lluis Alcanyis Hospital, Xàtiva, Valencia
  - Universitat de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sansone V, Maiorano E, Galluzzo A, Pascale V. Calcific tendinopathy of the shoulder: clinical perspectives into the mechanisms, pathogenesis, and treatment. Orthop Res Rev. 2018 Oct 3;10:63-72. doi: 10.2147/ORR.S138225. eCollection 2018. PMID 30774461
- [Result] Simpson M, Pizzari T, Cook T, Wildman S, Lewis J. Effectiveness of non-surgical interventions for rotator cuff calcific tendinopathy: A systematic review. J Rehabil Med. 2020 Oct 31;52(10):jrm00119. doi: 10.2340/16501977-2725. PMID 32830280
- [Result] Harvie P, Pollard TC, Carr AJ. Calcific tendinitis: natural history and association with endocrine disorders. J Shoulder Elbow Surg. 2007 Mar-Apr;16(2):169-73. doi: 10.1016/j.jse.2006.06.007. Epub 2006 Dec 22. PMID 17188907
- [Result] Louwerens JK, Sierevelt IN, van Hove RP, van den Bekerom MP, van Noort A. Prevalence of calcific deposits within the rotator cuff tendons in adults with and without subacromial pain syndrome: clinical and radiologic analysis of 1219 patients. J Shoulder Elbow Surg. 2015 Oct;24(10):1588-93. doi: 10.1016/j.jse.2015.02.024. Epub 2015 Apr 11. PMID 25870115
- [Result] Uhthoff HK, Loehr JW. Calcific Tendinopathy of the Rotator Cuff: Pathogenesis, Diagnosis, and Management. J Am Acad Orthop Surg. 1997 Jul;5(4):183-191. doi: 10.5435/00124635-199707000-00001. PMID 10797220
- [Result] Ioppolo F, Tattoli M, Di Sante L, Attanasi C, Venditto T, Servidio M, Cacchio A, Santilli V. Extracorporeal shock-wave therapy for supraspinatus calcifying tendinitis: a randomized clinical trial comparing two different energy levels. Phys Ther. 2012 Nov;92(11):1376-85. doi: 10.2522/ptj.20110252. Epub 2012 Jun 28. PMID 22745199
- [Result] Lafrance S, Doiron-Cadrin P, Saulnier M, Lamontagne M, Bureau NJ, Dyer JO, Roy JS, Desmeules F. Is ultrasound-guided lavage an effective intervention for rotator cuff calcific tendinopathy? A systematic review with a meta-analysis of randomised controlled trials. BMJ Open Sport Exerc Med. 2019 Mar 9;5(1):e000506. doi: 10.1136/bmjsem-2018-000506. eCollection 2019. PMID 31191964
- [Derived] Caballero I, Duenas L, Balasch-Bernat M, Fernandez-Matias R, Breso-Parra L, Gallego-Terres C, Aroca Navarro JE, Navarro-Bosch M, Lewis J, Lluch Girbes E. Effectiveness of non-surgical management in rotator cuff calcific tendinopathy (the effect trial): protocol for a randomised clinical trial. BMJ Open. 2024 Jan 4;14(1):e074949. doi: 10.1136/bmjopen-2023-074949. PMID 38176875